CLINICAL TRIAL: NCT03066726
Title: Does the Cerebroplacental Ratio (CPR) Predict Adverse Outcomes in Low Risk Pregnancies?
Acronym: CPR
Status: Terminated | Type: Observational
Why Stopped: Unable to meet recruitment target
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Virtua Medical Group (Other); Columbia University (Other); Saint Peters University Hospital (Other); Winthrop University Hospital (Other); New York Presbyterian Queens (Unknown)
Responsible Party: Principal Investigator, Todd Rosen, MD, Director, Maternal-Fetal Medicine, Rutgers, The State University of New Jersey
Other Study IDs: RU10312017
Record Dates: First submitted 2017-02-08; First posted 2017-02-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cerebroplacental Ratio
Keywords: Biophysical profile; Cesarean section; Estimated fetal weight; Middle cerebral artery; Umbilical artery; Fetal growth restriction; Pulsatility index; Estimated gestational age; Doppler
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPR less than the 10%le: Group of patients with fetuses with cerebroplacental ratio less than 10%le
- CPR greater or equal than 10%le: Group of patients with fetuses with cerebroplacental ratio greater or equal than 10%le

SUMMARY:
Ultrasound Doppler studies are used during pregnancy to help manage pregnancies complicated by fetal growth restriction. The cerebroplacental ratio may predict adverse outcomes in low risk pregnancies. In a prospective study, the investigators will examine whether fetuses with an abnormal CPR at or near term are at increased risk for being delivered by cesarean,

DETAILED DESCRIPTION:
This is a multicenter prospective study of low-risk nulliparous women who will be recruited if they are having an ultrasound at 36 weeks of estimated gestational age or greater. As part of the study, women will have umbilical and middle cerebral artery Doppler studies and the CPR will be calculated by dividing the middle cerebral artery PI by the umbilical artery PI. Providers caring for study subjects will be blinded to this result. Pregnancy outcomes in women with CPR values less than the 10th percentile for gestational age will be compared to those with CPR values above the 10th percentile.

A secondary aim of the study is to analyze CPR as a continuous variable.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant women between the ages of 18 and 45 years with low risk pregnancies who present for obstetrical ultrasound at 36 weeks of gestation or later with a planned delivery at a Perinatal Research Consortium hospital.

Exclusion Criteria:

* Multifetal pregnancy at the time of presentation
* Known fetal chromosomal anomaly
* Known fetal malformation
* Preeclampsia
* Fetal growth restriction
* Multiparity
* Prior cesarean section
* Placental abnormalities such as previa or accreta
* Pregestational diabetes
* Plan to deliver outside the Perinatal Research Consortium affiliated hospitals

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This is a multicenter prospective study of low-risk nulliparous women who will be recruited if they are having an ultrasound at 36 weeks EGA or greater.
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Cesarean delivery | From labor to delivery
  Cesarean delivery rate for non reassuring fetal heart tracings

SECONDARY OUTCOMES:
Total cesarean section rate | From labor to delivery
  Cesarean delivery rate for other indications other than non reassuring fetal heart tracings
Cord blood gases | At the time of delivery
  If obtained by the provider, umbilical (arterial or venous) cord pH
Cases of small for gestational age undetected prenatally | At time of delivery
  Neonates that were small for gestational age at time of delivery but were not detected prenatally
Birthweight/ birthweight percentile | At time of delivery
  Neonate birth weight and percentiles according to established weight charts will be recorded
Incidence of category 2 or 3 tracings | During labor
  As defined by the National Institutes of Health-National Institute of Child Health and Human Development Fetal Heart Tracings definitions and classifications
Distribution of CPR by estimated fetal weight | Measured during ultrasound between 36 weeks gestational age and delivery of the pregnancy.
  We will assess whether there is an association between the CPR and sonographic estimation of fetal weight.
Rate of operative vaginal delivery | At time of delivery
  Vaginal deliveries needing forceps or vacuum assistance
Neonatal Intensive Care Unit admission | Up to 28 days from delivery of the pregnancy
  Percentage of neonates admitted to the neonatal intensive care unit
Apgar scores at 1 and 5 minute | Scores assigned at 1 and 5 minutes of life by clinical staff.
  Standard assessment tool applied to all neonates in participating centers by clinical staff
Composite neonatal outcome | Up to 28 days from delivery of the pregnancy.
  The investigators will record a composite neonatal outcome including-respiratory distress, apnea, infection, hypoglycemia, hyperbilirubinemia, hypothermia, neurologic complication and neonatal death.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Rosen, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (6):
- United States (6):
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - Saint Peters University Hospital, New Brunswick, New Jersey
  - Virtua Medical Group, Sewell, New Jersey
  - New York Presbyterian-Queens Hospital, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prior T, Mullins E, Bennett P, Kumar S. Prediction of intrapartum fetal compromise using the cerebroumbilical ratio: a prospective observational study. Am J Obstet Gynecol. 2013 Feb;208(2):124.e1-6. doi: 10.1016/j.ajog.2012.11.016. Epub 2012 Nov 15. PMID 23159689
- [Background] Figueras F, Savchev S, Triunfo S, Crovetto F, Gratacos E. An integrated model with classification criteria to predict small-for-gestational-age fetuses at risk of adverse perinatal outcome. Ultrasound Obstet Gynecol. 2015 Mar;45(3):279-85. doi: 10.1002/uog.14714. Epub 2015 Jan 27. PMID 25358519
- [Background] DeVore GR. The importance of the cerebroplacental ratio in the evaluation of fetal well-being in SGA and AGA fetuses. Am J Obstet Gynecol. 2015 Jul;213(1):5-15. doi: 10.1016/j.ajog.2015.05.024. PMID 26113227
- [Result] Morales-Rosello J, Khalil A, Morlando M, Papageorghiou A, Bhide A, Thilaganathan B. Changes in fetal Doppler indices as a marker of failure to reach growth potential at term. Ultrasound Obstet Gynecol. 2014 Mar;43(3):303-10. doi: 10.1002/uog.13319. PMID 24488879